CLINICAL TRIAL: NCT04930965
Title: Louisiana Community-Engagement Alliance Against COVID-19 Disparities (LA-CEAL): Impact of HALT COVID Ambassador Program on Likelihood to Vaccinate
Brief Title: Impact of LA-CEAL HALT COVID-19 Ambassador Program on Likelihood to Vaccinate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1600; OT2 HL158260 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-06-18 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Covid19; Vaccine Refusal
Keywords: Community Health Worker
MeSH Terms: conditions — COVID-19; Vaccination Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Community health worker engagement
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Community health worker engagement — 3-4 in-person or virtual engagements (individual or group sessions) over 1 month, each engagement lasting 30 minutes to 1 hour
  Arms: Intervention

SUMMARY:
The purpose of the study is to assess the effectiveness of the HALT COVID Ambassador educational outreach program on increasing likelihood to vaccinate against COVID-19

DETAILED DESCRIPTION:
Investigators will use a randomized controlled trial to test the effectiveness of HALT COVID educational outreach by HALT COVID Ambassadors. HALT COVID Ambassadors will receive training to answer common vaccine questions & address misconceptions; conduct motivational interviewing; and implement basic behavioral economics and related strategies to remove barriers to vaccination. A random sample of FQHC patients will be identified in EHR data downloads of adult patients seen in the last year and contacted by telephone to gain consent and assess eligibility. A total of 100 individuals will be enrolled into the trial and randomized to intervention (engagement with the HALT COVID Ambassador over a 1 month period via in-person or virtual sessions exploring their own questions and concerns about vaccines) or usual care (no extra engagement). Baseline, 1-month, and 2-month follow-up surveys will assess for vaccine likelihood.

ELIGIBILITY:
Inclusion Criteria:

* Unlikely to vaccinate in next month
* Age >=18 years
* Self-identification as Black or African American
* Ability to understand and speak English
* Willingness to engage with HALT COVID Ambassador via in-person or virtual sessions exploring questions and concerns about vaccines

Exclusion Criteria:

* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: No intervention
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 27 | 29
Completed | 20 | 24
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.4) | 44.1 (13.4) | 42.7 (13.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 6 | 8 | 14
  Women | 21 | 21 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 29 | 53
  White | 0 | 0 | 0
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Difference in Proportion of Participants "Likely to Vaccinate" Between Study Arms at Month 1
Description: Vaccine likelihood will be measured using a single question adapted from the CEAL Common Survey (i.e., "On a scale from 1 to 7, with 1 being 'not at all likely' and 7 being 'very likely', how likely are you to get a COVID-19 vaccine in the next month?"), with "likely to vaccinate" defined as a score of 5-7.
Time Frame: Month 1 follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 21 | 26
Participants | 1 | 3

2. Secondary Outcome: Difference in Proportion of Participants "Likely to Vaccinate" Between Study Arms at Month 2
Description: as for outcome 1
Time Frame: Month 2 follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 24
Participants | 4 | 4

3. Secondary Outcome: Difference in Proportion of Participants Who Have Received >=1 Dose of Vaccine Between Study Arms at Month 1
Description: Receipt of vaccination will be measured by self-report
Time Frame: Month 1 follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 21 | 26
Participants | 1 | 2

4. Secondary Outcome: Difference in Proportion of Participants Who Have Received >=1 Dose of Vaccine Between Study Arms at Month 2
Description: Receipt of vaccination will be measured by self-report
Time Frame: Month 2 follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 24
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04930965/Prot_SAP_000.pdf